CLINICAL TRIAL: NCT00042952
Title: A Phase II Study Of Imatinib Mesylate (Gleevec, Formerly Known As STI571; IND 61,135, NSC #716051) In Patients With Refractory Seminoma
Brief Title: Imatinib Mesylate in Treating Patients With Progressive, Refractory, or Recurrent Stage II or Stage III Testicular or Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02481; CLB-90105; U10CA031946 (NIH); CDR0000069487 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Ovarian Dysgerminoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Ovarian Germ Cell Tumor; Stage II Malignant Testicular Germ Cell Tumor; Stage II Ovarian Germ Cell Tumor; Stage III Malignant Testicular Germ Cell Tumor; Stage III Ovarian Germ Cell Tumor; Testicular Seminoma
MeSH Terms: conditions — Dysgerminoma; Testicular Neoplasms; Seminoma | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate and surgical resection) (Experimental): Patients receive oral imatinib mesylate once daily. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients who achieve a partial response or stable disease with normalization of human chorionic gonadotropin may undergo surgical resection of residual lesions at each tumor status assessment. If residual viable germ cell tumor is present in the resected specimen, patients may resume imatinib mesylate. If no viable germ cell tumor is present in the resected specimen, then no further therapy is administered.
  Interventions: Drug: imatinib mesylate; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Procedure: therapeutic conventional surgery — Undergo surgical resection
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have progressive, refractory, or recurrent stage II or stage III testicular cancer or stage II or stage III ovarian cancer following cisplatin-based chemotherapy

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the activity of imatinib mesylate in patients with progressive, refractory, or recurrent pure testicular seminoma or ovarian germ cell dysgerminoma after cisplatin-based chemotherapy.

II. Determine the toxicity of this drug in this patient population. III. Determine KIT expression and identify mutations in the c-kit gene in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate once daily. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients who achieve a partial response or stable disease with normalization of human chorionic gonadotropin may undergo surgical resection of residual lesions at each tumor status assessment. If residual viable germ cell tumor is present in the resected specimen, patients may resume imatinib mesylate. If no viable germ cell tumor is present in the resected specimen, then no further therapy is administered.

Patients are followed every 3 months for 1 year and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study within 32-38 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pure testicular seminoma or ovarian germ cell dysgerminoma

  * Histologic documentation of metastatic/recurrent disease not required
* Alpha-fetoprotein level must be normal, unless abnormal level is explained by other conditions and approved by the study chair
* Clinical stage II or III
* Progressive, refractory, or recurrent disease, meeting at least 1 of the following criteria:

  * Measurable progressive disease
  * Biopsy-proven residual disease
  * Persistently elevated or rising B-human chorionic gonadotropin (HCG) titers, defined as at least 2 values above the upper limit of normal (ULN)
* Cisplatin-refractory disease without option of potentially curative therapy, meeting 1 of the following criteria:

  * Failed high-dose chemotherapy with peripheral blood stem cell transplantation (PBSCT) or autologous bone marrow transplantation (AuBMT)
  * Ineligible for or refused PBSCT or AuBMT
  * Unlikely to achieve long-term benefit from PBSCT or AuBMT
* Current evidence of metastatic disease

  * Unidimensionally measurable target lesions

    * At least 20 mm by conventional techniques (e.g., physical examination for clinically palpable lymph nodes and superficial skin lesions or chest x-ray for clearly defined lung lesions surrounded by aerated lung)
    * At least 10 mm by spiral CT scan or MRI
    * If measurable disease is confined to a solitary lesion, then its neoplastic nature must be confirmed by histology
    * Ultrasound may not be used to measure tumor lesions that are not easily accessible clinically
* Non-measurable/non-target lesions, with HCG at least ULN, including the following:

  * Bone lesions
  * Pleural or pericardial effusions
  * Ascites
  * CNS lesions
  * Leptomeningeal disease
  * Irradiated lesions, unless progression documented after radiotherapy
* Performance status - ECOG 0-2
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL (transfusion allowed)
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No other severe and/or uncontrolled concurrent medical illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* See Disease Characteristics
* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy
* No concurrent hormonal therapy except steroids for adrenal failure, hormones for non-disease-related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* Prior radiotherapy to a symptomatic lesion or one that may produce disability (e.g., unstable femur) allowed
* No concurrent palliative radiotherapy
* No concurrent grapefruit juice
* No concurrent warfarin for therapeutic anticoagulation (concurrent mini-dose warfarin [1 mg orally per day] as prophylaxis allowed)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-06; Primary Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Response rate defined as either a complete or partial response using RECIST criteria | Up to 2 years
  Response rate (CR+PR) and exact 95% confidence interval based on the binomial distribution for the response rate will be computed.

SECONDARY OUTCOMES:
Grade 1 or higher toxicities assessed using CTC)version 2 | Up to 2 years
  Toxicities will be tabulated.
Duration of response | From first response (CR or PR) to the date of disease progression or death, assessed up to 2 years
  The Kaplan-Meier product-limit method will be used.
Disease-free survival | From the date of initiation of treatment to date of progression or death due to any cause, whichever occurs first, assessed up to 2 years
  The Kaplan-Meier product-limit method will be used.
Overall survival | From date of initiation of treatment to date of death due to any cause, assessed up to 2 years
  The Kaplan-Meier product-limit method will be used.
Proportion of patients with mutations in the c-KIT gene | Up to 2 years
  The 95% confidence interval will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ryan, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States